CLINICAL TRIAL: NCT01474668
Title: A Phase I Study to Investigate the Absorption, Metabolism, and Excretion of [14c]-GDC-0941 Following Single Oral Dose Administration in Healthy Male Subjects
Brief Title: Study to Investigate the Absorption, Metabolism, and Excretion of [14C]-GDC-0941 Following Single Oral Dose Administration in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GP27917
Record Dates: First submitted 2011-11-16; First posted 2011-11-18 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — 2-(1H-indazol-4-yl)-6-(4-methanesulfonylpiperazin-1-ylmethyl)-4-morpholin-4-ylthieno(3,2-d)pyrimidine

ARMS (1):
- A (Experimental): Experimental
  Interventions: Drug: GDC-0941

INTERVENTIONS:
Drug: GDC-0941 — Single oral dose\n \n\n\n\n

SUMMARY:
This study will be an open-label, non-randomized, absorption, metabolism, and excretion study of [14C]-GDC 0941 administered as an oral dose to 6 healthy male subjects following at least a 10-hour fast from food (not including water).

ELIGIBILITY:
Inclusion Criteria:

* Within BMI range 18.5 to 29.9 kg/m2, inclusive
* In good health, determined by no clinically significant findings from medical history, 12-lead ECG, and vital signs
* Clinical laboratory evaluations within the reference range for the test laboratory
* Negative test for selected drugs of abuse at Screening and at Check-in
* Negative hepatitis panel (including hepatitis B surface antigen [HBsAg], hepatitis C virus antibody [anti-HCV]) and negative HIV antibody screens
* Subjects will either be sterile or agree to use an approved form of contraception from Check-in until 45 days following Study Completion/ET
* Agree not to donate sperm from Screening throughout the study period and for at least 3 months (90 days) after the last dose of study drug
* A minimum of 1 to 2 bowel movements per day

Exclusion Criteria:

* Significant history or clinical manifestation of any significant metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, or psychiatric disorder
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance
* History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs (except that appendectomy and hernia repair will be allowed)
* History of Gilbert's Syndrome
* History of diabetes mellitus and/or elevated fasting glucose at baseline
* History or presence of an abnormal ECG
* History of alcoholism or drug addiction within 1 year prior to Check-in
* Participation in more than one other radiolabeled investigational study drug trial within 12 months prior to Check-in. The previous radiolabeled study drug must have been received more than 6 months prior to Check-in for this study and the total exposure from this study and the previous study will be within the recommended levels considered safe
* Exposure to significant radiation within 12 months prior to Check-in
* Use of any tobacco-containing or nicotine-containing products within 6 months prior to Check-in or positive urine drug screen for cotinine
* Participation in any other investigational study drug trial in which receipt of an investigational study drug occurred within 5 half-lives or 30 days, whichever is longer, prior to Check-in
* Use of any prescription medications/products within 14 days prior to Check-in, unless deemed acceptable by the Investigator
* Use of any over-the-counter (OTC), non-prescription preparations (including vitamins, minerals, and phytotherapeutic/herbal/plant derived preparations) within 7 days prior to Check-in
* Use of alcohol-, grapefruit-, or caffeine-containing foods or beverages within 72 hours prior to Check-in, unless deemed acceptable by the Investigator
* Poor peripheral venous access
* Donation of blood from 30 days prior to Screening or of plasma from 2 weeks prior to Screening
* Receipt of blood products within 2 months prior to Check-in
* Any acute or chronic condition that, in the opinion of the Investigator, would limit the subject's ability to complete and/or participate in this clinical study

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2011-10; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic property based on the plasma concentrations of total radioactivity and GDC-0941: apparent terminal elimination half-life | up to approximately 6 weeks or early study discontinuation
Pharmacokinetic property based on the plasma concentrations of total radioactivity and GDC-0941: apparent terminal phase elimination rate constant | up to approximately 6 weeks or early study discontinuation
Pharmacokinetic property based on the plasma concentrations of total radioactivity and GDC-0941: apparent total clearance | up to approximately 6 weeks or early study discontinuation
Pharmacokinetic property based on the plasma concentrations of total radioactivity and GDC-0941: apparent volume of distribution | up to approximately 6 weeks or early study discontinuation
Pharmacokinetic property based on the plasma concentrations of total radioactivity and GDC-0941: area under the concentration-time curve extrapolated to infinity | up to approximately 6 weeks or early study discontinuation
Pharmacokinetic property based on the plasma concentrations of total radioactivity and GDC-0941: area under the concentration-time curve from Hour 0 to the last measurable concentration | up to approximately 6 weeks or early study discontinuation
Pharmacokinetic property based on the plasma concentrations of total radioactivity and GDC-0941: maximum observed concentration | up to approximately 6 weeks or early study discontinuation
Pharmacokinetic property based on the plasma concentrations of total radioactivity and GDC-0941: time to maximum concentration | up to approximately 6 weeks or early study discontinuation

SECONDARY OUTCOMES:
Amount of drug excreted in the feces over the sampling interval | up to approximately 6 weeks or early study discontinuation
Percent excreted in feces | up to approximately 6 weeks or early study discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Scott Holden, M.D., Study Director — Genentech, Inc.
Locations (1):
- Madison, Wisconsin, United States